CLINICAL TRIAL: NCT07355205
Title: A Phase II, Single-Center, Open-Label Study of First-Line Ipilimumab Plus Nivolumab and Nogapendekin Alfa Inbakicept (N-803) in Patients With Stage IV or Recurrent Non-Small Cell Lung Cancer (FLINN)
Brief Title: First-Line Ipilimumab Plus Nivolumab and Nogapendekin Alfa Inbakicept (N-803) in Patients With Stage IV or Recurrent Non-Small Cell Lung Cancer
Acronym: FLINN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: ImmunityBio, Inc. (Industry); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-X396
Record Dates: First submitted 2026-01-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer Stage IV; Non-small Cell Lung Cancer Recurrent
Keywords: Non-small cell lung cancer; Stage IV; Immunotherapy; IL-15 super agnoist
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Nivolumab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ipilimumab plus Nivolumab and Nogapendekin alfa inbakicept (N-803) (Experimental): Consenting and eligible patients will receive nivolumab intravenously (IV) on Days 1 and 22, ipilimumab IV on Day 1, and nogapendekin alfa inbakicept subcutaneously (SC) on Days 1 and 22 of each cycle for Cycles 1 through 4; ipilimumab will be discontinued after Cycle 4 and patients will continue to receive nivolumab and nogapendekin alfa inbakicept on the same schedule for up to 2 years. Cycles are 42 days (6 weeks).
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Nogapendekin alfa inbakicept

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab will be given intravenously at a dose of 1mg/kg.
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab will be given intravenously at a dose of 360mg.
  Other Names: Opdivo
Drug: Nogapendekin alfa inbakicept — Nogapendekin alfa inbakicept will be given subcutaneously at a dose of 15 μg/kg.
  Other Names: N-803; Anktiva

SUMMARY:
This is an open-label, single center, one cohort, non-randomized, phase II study. The aim of the study is to evaluate the efficacy and safety of the combination of nivolumab and ipilimumab with nogapendekin alfa inbakicept in patients with stage IV or recurrent non-small cell lung cancer (NSCLC). It is hypothesized that the study treatment will be safe and well tolerated and will improve progression-free survival when compared to a historical study which treated advanced NSCLC patients with nivolumab plus ipilimumab. Patients will be treated in cycles lasting 6 weeks with two to three different chemotherapy drugs to up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, previously untreated or recurrent metastatic NSCLC.
* Availability of archival biopsy tissue or willingness to undergo a biopsy prior to C1D1 for biomarker analysis, including PD-L1 by IHC using a CLIA-certified test. Results of the PD-L1 testing are not required for enrollment.
* Measurable disease per RECIST 1.1.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Adequate organ and marrow function, as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN without hepatic metastasis and ≤ 5 x IULN with hepatic metastasis
  * Total bilirubin ≤ 2 x IULN (except participants with Gilbert's syndrome who must have total bilirubin < 3.0 mg/dL)
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
  * INR ≤ 1.5 unless using therapeutic anticoagulation
  * PTT/aPTT < 1.5 x IULN unless using therapeutic anticoagulation
* Patients with brain metastases are eligible if they have previously treated with surgery or radiation therapy, are neurologically stable after a washout period of at least 2 weeks, and are not receiving corticosteroids at dose higher than 10 mg of prednisone or equivalent on C1D1.
* The effects of the treatment regimen on the developing human fetus are unknown. For this reason, people of childbearing potential and people able to father a child must agree to use highly effective methods of contraception, according to the protocol, from the time of consent through 6 months after the last dose of study treatment.
* Ability to understand and willingness to sign an IRB-approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Mixed histology including small cell lung cancer.
* Tumor harboring EGFR mutation, HER2 mutation, ALK fusion, ROS1 fusion or RET fusion.
* Use of any live vaccines within 28 days of C1D1.
* Prior chemotherapy in the adjuvant setting or during concurrent radiation therapy for locally advanced disease within 12 months prior to enrollment. If the interval from the last treatment is 12 months or longer, the patient is eligible.
* Radiation therapy within 14 days prior to C1D1.
* History of major surgery within 14 days prior to C1D1.
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study treatment hazardous, including but not limited to:

  * History of interstitial lung disease or noninfectious pneumonitis,
  * Active viral, bacterial or fungal infections requiring parenteral treatment within 14 days of C1D1,
  * Clinically significant cardiovascular disease,
  * A condition that may obscure the interpretation of toxicity determination or AEs,
  * History of prior solid-organ transplantation.
* Concurrent medical condition requiring the use of supra-physiologic doses of corticosteroids (> 10 mg/day of oral prednisone or equivalent) or immunosuppressive medications (absorbable topical corticosteroids are not excluded).
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing not required in the absence of known history of infection.
* Evidence of chronic hepatitis B (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing not required in the absence of known history of infection.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy.

  * Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
  * Participants with asthma who require intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections will not be excluded from this study.
  * Participants on chronic systemic corticosteroids will be excluded from the study.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of C1D1.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any agents used in the study, or known hypersensitivity to recombinant proteins, or any excipient contained in the trial formulations.
* Pregnant and/or breastfeeding. People of childbearing potential must have a negative pregnancy test within 7 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Start of treatment through 2 years after end of treatment (up to 4 years)
  PFS is defined as the duration of time from the start date of study treatment to the date of earliest progression or death, whichever occurs first. Patients who neither progress nor die by the data cutoff date will be censored at the last follow up date.

SECONDARY OUTCOMES:
Adverse event effect rate | Start of treatment through 100 days after discontinuation of therapy (up to 2 years and 100 days)
  Defined as the number of study treatment related adverse events (AEs) and discontinuations due to treatment-related AEs. Adverse events will be assessed using the CTCAE v5.0 criteria.
Disease control rate (DCR) | Start of treatment through 2 years after end of treatment (up to 4 years)
  DCR is defined as the proportion of patients achieving either a complete response (CR), partial response (PR), or stable disease (SD), according to RECIST 1.1.
  Complete Response (CR): Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Duration of response (DoR) | Start of treatment through 2 years after end of treatment (up to 4 years)
  DoR is defined as the time from the confirmation of a CR of PR according to RECIST 1.1 until the first date that recurrent or progressive disease is objectively documented or death from any cause.
  Complete Response (CR): Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Objective response rate (ORR) | Start of treatment through completion of treatment or progression (up to 2 years)
  ORR is defined as the proportion of patients achieving CR or PR measured according to RECIST 1.1.
  Complete Response (CR): Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Immune-related best overall response (iBOR) | Start of study treatment to up to 2 years after the end of treatment (up to 4 years)
  iBOR is defined as the proportion of the best confirmed immune-related response recorded from the start of the study treatment until disease progression, the end of treatment, or death, whichever comes first, according to iRECIST guideline.
Immune-related progression-free survival (iPFS) | Start of study treatment up to 2 years after treatment is completed (up to 4 years)
  iPFS is defined as the time from the start date of study treatment to date of confirmed immune-related progressive disease by investigator's assessment or death from any cause, whichever occurs first.
  Immune unconfirmed progressive disease (iUPD) is defined according to iRECIST guidelines.
Overall survival (OS) | Start of study treatment up to 2 years after treatment is completed (total 4 years)
  OS is defined as the duration of time from the start date of study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Giordano Fabricio Cittolin Santos, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu